CLINICAL TRIAL: NCT03364322
Title: Prospective Study for Influencing Factors on Dry Eye Syndrome, Ocular Surface Disease and Treatment
Brief Title: Influencing Factors on Dry Eye Syndrome and Ocular Surface Disease
Status: Completed | Type: Observational
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Young Joo Shin, Principal Investigator, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: 2016-06-73
Record Dates: First submitted 2017-11-25; First posted 2017-12-06 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Dry Eye Syndrome; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dry eye syndrome
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
Dry eye syndrome and ocular surface disease are very important ophthalmologic diseases. It is known that various inducers are involved. However, it is still necessary to study how influencing factors are related to dry eye syndrome and ocular surface disease and how treatment for dry eye syndrome and ocular surface disease is helpful.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ocular discomfort related to DED who visit the Hallym University Kangnam Sacred Heart Hospital between June 2016 and June 2017.

Exclusion Criteria:

* Subjects who are elderly (≥80 years old) or have an autoimmune disease (e.g., Sjögren's syndrome and systemic lupus erythematosus) are excluded.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ocular discomfort related to DED who visit the Hallym University Kangnam Sacred Heart Hospital between June 2016 and June 2017.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Ocular surface disease index | 1 day
  The ocular surface disease index survey in completed at the time of the exam. This scale ranges from 0 to 100 higher scores representing greater disability.

SECONDARY OUTCOMES:
Tear break-up time | 1 day
Schirmer tear secretion test | 1 day
  Schirmer tear secretion test (mm) without anesthesia was performed using strip (Color Bar; Eagle vision. Memphis, TN)
Corneal fluorescence staining | 1 day
  Corneal staining with fluorescein solution is graded at the time of the exam on a scale of 0 to 5 using the oxford scoring system with 5 being the most severe staining.

OTHER OUTCOMES:
Tear osmolarity | 1 day
  The tear film osmolarity (mOsm) is measured using TearLab (TearLab Co., San Diego, CA).
Eyelid hyperemia | 1 day
  Graded as follows. 0=none, 1= mild, 2=mod, and 3=severe
Conjunctivochalasis | 1 day
  Graded as follows. 0=none, 1= mild, 2=mod, and 3=severe fixed fold
visual analogue pain score | 1 day
  visual analogue pain score indicates a higher level of discomfort. 0 to 10.
modification of SPEED score | 1 day
  SPEED score using questionnaire indicates a higher level of discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sacred Heart Hospital, Seoul, South Korea